CLINICAL TRIAL: NCT00418015
Title: Mu-Opioid Receptor Genetic Polymorphism and the Duration of Intrathecal Fentanyl Labor Analgesia. Mu-Opioid Receptor Genetic Polymorphism and the Efficacy of Postoperative Intrathecal Morphine Analgesia
Brief Title: Mu-Opioid Receptor Genetic Polymorphism and Intrathecal Analgesia
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Other Study IDs: 0524-025
Record Dates: First submitted 2006-12-31; First posted 2007-01-04 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Labor Pain; Post-cesarean Delivery
Keywords: µ-opioid receptor; neuraxial labor analgesia; pharmacogenetics
MeSH Terms: conditions — Labor Pain | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Labor analgesia: Labor analgesia receiving fentanyl labor analgesia
  Interventions: Procedure: Blood Draw
- Cesarean delivery analgesia: Cesarean delivery analgesia consisting of spinal fentanyl and morphine
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Blood for OPRM1 analysis

SUMMARY:
Pharmacogenetics has allowed clinicians to identify associations between an individual's genetic profile and his/her response to drugs. The A118G (c.188A>G)is a single nucleotide polymorphism (SNP) of the mu-opioid receptor (OPRM1). The mutated protein, N40D, appears to increase the binding affinity and potency of beta-endorphin approximately 3-fold. Individuals carrying the variant receptor gene (A118G) may show differences in some of the functions mediated by beta-endorphin action at the altered OPRM1. Combined spinal-epidural (CSE) analgesia is a commonly utilized technique for labor analgesia. Analgesia is initiated with the intrathecal administration of a lipid-soluble opioid (e.g. fentanyl), sometimes combined with a local anesthetic. The mean (± SD) duration of analgesia after intrathecal fentanyl 25 microgram was 89 ± 43 min. The ED50 of intrathecal fentanyl for labor analgesia varies between 14 microgram to 18.2 microgram. The wide variability in the duration of analgesia, as was well the differences in ED50 may result from differences known to affect labor pain (e.g., ethnicity, parity, stage of labor). Another possible explanation for the differences in opioid requirements and duration, as well as incidence of side effects such as itching and nausea/vomiting, is that opioid responsiveness is determined by genetic variability of the µ-opioid receptor. The ED50 for intrathecal fentanyl labor analgesia was significantly lower for parturients carrying the A118G variant of the mu-opioid receptor, compared to parturients with the A118 wild type receptor. The purpose of this study is to determine whether polymorphism at nucleotide 118 of OPRM1 influences the duration of intrathecal opioid (fentanyl) labor analgesia, and intrathecal opioid (morphine) postoperative analgesia.

DETAILED DESCRIPTION:
Study 1 (intrathecal fentanyl): The primary outcome variable is duration of intrathecal fentanyl analgesia. A two-sided log rank test with an overall sample size of 152 subjects (wild type OPRM1 = 106, variant OPRM1 = 46) achieves 80% power at α = 0.05 to detect a difference of 0.2 between 0.5 and 0.3 (the proportion of subjects with continuing intrathecal fentanyl analgesia after 70 min). This assumes that 70% of subjects will have the wild-type MUOR1 phenotype, and 30% the variant phenotype. To account for anticipated subject dropout, 175 subjects will be enrolled in the study.

Study 2 (intrathecal morphine): The primary outcome variable is amount of rescue analgesia (morphine equivalents) necessary for 24 h after the intrathecal morphine injection. An overall sample size of 71 subjects (wild type OPRM1 = 50, variant OPRM1 = 21) achieves 81% power to detect a difference of 15 mg morphine equivalents between the null hypothesis that both group means are 40 mg morphine equivalents and the alternative hypothesis that the mean of one group is 25 mg morphine equivalents. The estimated group standard deviations are 20 mg morphine equivalents with alpha = 0.05 using a two-side Mann-Whitney test assuming that the actual distribution is uniform. This assumes that 70% of subjects will have the wild-type OPRM1 phenotype, and 30% the variant phenotype. To account for anticipated subject dropout, 90 subjects will be enrolled in the study.

Protocol specific methods:

Study 1: Eligible parturients admitted to the Labor and Delivery Unit of Prentice Women's Hospital will be approached for study participation immediately after the routine preanesthetic evaluation. This occurs shortly after admission to the Labor and Delivery Unit. Women who agree to participate will give written, informed consent at this time.

Venous blood will be obtained for genetic analysis of the 118 position of the µ-opioid receptor gene shortly after the subject consents to study participation, either through an intravenous catheter placed for routine intravenous access for labor and delivery, or through a fresh venipuncture. A total of 10 mL blood will be collected into two 5 mL EDTA tubes. The tubes will be batched, coded and stored in a 40C refrigerator until they will be send (1x/month) to the laboratory of Dr. J. L. Blouin, care of Dr. Landau, at the Hopitaux Universitaires de Geneve. Genetic analysis will be performed as described below. When the subject first requests analgesia, her cervix will be examined (this is routine procedure prior to initiating analgesia). If the cervix is dilated between 2 and 5 cm, the parturient will be included in the study. Visual analogue score (VAS) for pain (100 mm line where 0 mm = no pain and 100 mm = worst possible pain) will be determined immediately before initiation of analgesia. Combined spinal-epidural analgesia will be initiated in the sitting position per routine with intrathecal fentanyl 25 microgram. An epidural catheter will be sited. No drug will be injected through the epidural catheter until the parturient requests analgesia again. The parturient will be placed in the lateral position after the epidural catheter is secured. A VAS will be determined 10 min after the intrathecal injection.

The primary outcome variable is duration of intrathecal fentanyl analgesia.At the time the parturient requests additional analgesia, the cervix will be examined. A VAS will be determined. In addition, the parturient will be asked about the presence of pruritus since the initiation of analgesia (none, mild, moderate, severe), nausea (none, mild, moderate or severe), and vomiting (yes, no). An epidural test dose will be administered (lidocaine 1.5% with epinephrine 1:200,000). Assuming a negative test dose, bupivacaine 0.125% will be injected incrementally to a T10 sensory level. Epidural analgesia will be maintained with patient controlled epidural analgesia (PCEA) (bupivacaine 0.0625% with fentanyl 1.95 micro grams/mL: background infusion 15 mL/h, PCEA bolus 5 mL, lockout 10 min, maximum 30 mL/h) as per routine.

The study ends after the parturient delivers and the epidural infusion is discontinued. At this time the subject will be asked about her satisfaction with labor analgesia (100 mm scale, 0 mm = not satisfied at all, 100 mm = very satisfied).

The following data will be collected: maternal age, height, weight, race (self-described), cervical dilation at initiation of analgesia, time and cervical dilation at 2nd request for analgesia, maximum oxytocin dose, time to complete cervical dilation (10 cm), time to delivery, mode of delivery, neonatal weight, Apgar scores and umbilical blood gas values (obtained as part of routine care), total dose of epidural bupivacaine and other local anesthetics, total dose of epidural fentanyl, number of PCEA boluses and number of manual boluses (by the anesthesiologist).

Cases will be excluded from data analysis if CSE analgesia is not performed, if there is no analgesia (VAS > 10 mm) 10 minutes after the intrathecal injection (failure of CSE technique), if cervical dilation is 8 cm within 60 minutes of intrathecal injection, or if the patient has a cesarean delivery. These cases will be reported.

Study 2: Eligible women admitted to the Labor and Delivery Unit of Prentice Women's Hospital for planned Cesarean delivery will be approached for study participation immediately after the routine preanesthetic evaluation. This occurs shortly after admission to the Labor and Delivery Unit. Women who agree to participate will give written, informed consent at this time.

Venous blood will be obtained for genetic analysis of the 118 position of the µ-opioid receptor gene shortly after the subject consents to study participation, either through an intravenous catheter placed for routine intravenous access for labor and delivery, or through a fresh venipuncture. A total of 10 mL blood will be collected into two 5 mL EDTA tubes. The tubes will be batched, coded and stored in a 4oC refrigerator until they are sent (1time/month) to the laboratory of Dr. J. L. Blouin, care of Dr. Landau, at the Hospitaux Universitaires de Geneve. Genetic analysis will be performed as described below Routine aspiration prophylaxis will be administered (intravenous ranitidine and metoclopramide, and oral antacid). Spinal anesthesia will be initiated in the sitting position in the routine manner with bupivacaine 12 mg (1.6 mL 0.75% hyperbaric bupivacaine), fentanyl 15 µg, and morphine 150 micrograms. Subjects will be placed in the supine left uterine displacement position immediately after the intrathecal injection. The level of cephalad sensory blockade will be determined 30 min after the intrathecal injection using von Frye hairs. Subjects with a sensory level below T6, or those that require intraoperative systemic opioid supplementation, will be excluded from further study participation.

In the PACU and for 24 hours after surgery, patients will receive ibuprofen 600 mg po q6h as per standard protocol. Patients may request rescue analgesia if they are experiencing discomfort. Rescue medication will consist of hydrocodone 10 mg plus acetaminophen 325 mg per os. An additional dose of hydrocodone 10 mg plus acetaminophen 325 mg will be provided after 1 hour if the pain is not relieved. These are routine oral analgesic medications for postoperative Cesarean delivery analgesia. Standard orders will be written for monitoring sedation and respiratory rate, and treatment of side effects (nausea, vomiting, pruritus and respiratory depression).

The primary outcome variable is amount of rescue morphine equivalent analgesia required for the 24 hours after the intrathecal morphine injection.18 The time of first rescue analgesia request will be noted, and the VAS will be determined at the time of request for rescue analgesia. In addition, the parturient will be asked to provide a VAS for pain at 4, 8, 12, 18, and 24 hours after the intrathecal injection. The presence of pruritus (none, mild, moderate, severe), nausea (none, mild, moderate or severe), and vomiting (yes, no) will be determined at 4 and 24 h after the intrathecal injection.

The study ends 24 h after the intrathecal injection. At this time the subject will be asked about her satisfaction with postoperative analgesia (100 mm scale, 0 mm = not satisfied at all, 100 mm = very satisfied). Further analgesia will not be dictated by study protocol.

The following data will be collected: maternal age, height, weight, race (self-described), requirement for supplemental intraoperative sedation, neonatal weight, intra- or postoperative treatment for pruritus, nausea or vomiting. In addition to the time to first request for supplemental oral analgesia, the following will be recorded: supplement analgesia dose requirements (number of acetaminophen/hydrocodone tablets) at 4, 8, 12, 18, and 24 h after the intrathecal injection.

DNA collection: Peripheral blood will be collected in 2 5ml EDTA tubes (total 10ml). DNA will be prepared by non-phenolic methods using Puregene Blood Extraction Kit (Gentra, Minneapolis, MN) and tested for molecular weight on gel electrophoresis and purity quality by optical densitometry measure (ratio 260/280 nm).

SNP genotyping: For identification of allelic distribution of the A118G SNP, 20-60 ng of DNA from individuals will be first amplified by PCR (on thermocycler apparatuses equipped with a 96 well-microtiter plate block) using primers designed in the vicinity of the SNPs. The SNP will be then genotyped in amplified products by minisequencing (Pyrosequencing).

Pyrosequencing: PCR using cDNA specific primers (spanning an intron in genomic DNA), in which the forward primer is labeled with 5' biotin is performed under standard conditions, and the product is analyzed by the Pyrosequencing method. Briefly, an internal primer is designed two nucleotides before the mutation site, so that the two mRNA populations could be assayed by quantifying the relative amounts of each allele present in the PCR product. DNA from normal and affected subjects are used as controls.

PCR products are immobilized with Dynabeads (Dynal, Oslo, Norway) by a 15 min, 65 oC incubation in a buffer containing 10mM Tris-HCl, 2M NaCl, 1mM EDTA and 0.1% Tween 20. PCR products are then removed from solution using magnetic separation, denatured with NaOH 0.5 M and washed with 200mM Tris-Acetate, 50mM MgAc2. The remaining single stranded DNA is then hybridized with the internal 'sequencing' primer, by heating the mix to 80oC, and slowly cooling it to room temperature. Next enzyme and substrate mixes are automatically added to each well, and the reactions proceed at 28oC, by the sequential addition of single nucleotides at a predetermined order. Luciferase peak heights are proportional to the number of nucleotide incorporations, which has been shown to be very quantitative (5% error rate) in a number of experimental settings.

Coded DNA samples will be stored in Dr. Blouin's laboratory. No further sequencing will be done unless subjects signed the consent form for further future studies.

ELIGIBILITY:
Inclusion Criteria:

Study 1: Laboring Women

* Nulliparous women in spontaneous labor or with spontaneous rupture of membranes
* Term pregnancy (≥ 37 weeks gestation)
* Vertex presentation
* Healthy, ASA PS 1-2
* Desire neuraxial labor analgesia.

Study 2: Cesarean Delivery

* Nulliparous women undergoing elective primary Cesarean delivery (e.g., for breech presentation, macrosomia)
* Term pregnancy (≥ 37 weeks gestation)
* Healthy, ASA PS 1-2
* Desired spinal anesthesia.

Exclusion Criteria:

Study 1: Laboring Women

* Chronic or pregnancy induced disease
* Chronic opioid use
* History of substance abuse
* Systemic opioid analgesia before initiation of neuraxial labor analgesia
* Cervical dilation < 2 cm or > 5 cm of time of request for neuraxial analgesia
* Allergy to fentanyl

Study 2: Cesarean delivery

* Chronic or pregnancy induced disease
* Chronic opioid use
* Previous abdominal or pelvic surgery
* Allergy to fentanyl, morphine, or bupivacaine
* BMI ≥ 40 kg/m2
* History of substance abuse
* Failed spinal anesthesia
* Requirement for systemic opioid supplementation during Cesarean delivery.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2005-10; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Wong, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Palmer SN, Giesecke NM, Body SC, Shernan SK, Fox AA, Collard CD. Pharmacogenetics of anesthetic and analgesic agents. Anesthesiology. 2005 Mar;102(3):663-71. doi: 10.1097/00000542-200503000-00028. PMID 15731608
- [Background] Befort K, Filliol D, Decaillot FM, Gaveriaux-Ruff C, Hoehe MR, Kieffer BL. A single nucleotide polymorphic mutation in the human mu-opioid receptor severely impairs receptor signaling. J Biol Chem. 2001 Feb 2;276(5):3130-7. doi: 10.1074/jbc.M006352200. Epub 2000 Nov 6. PMID 11067846
- [Background] Bond C, LaForge KS, Tian M, Melia D, Zhang S, Borg L, Gong J, Schluger J, Strong JA, Leal SM, Tischfield JA, Kreek MJ, Yu L. Single-nucleotide polymorphism in the human mu opioid receptor gene alters beta-endorphin binding and activity: possible implications for opiate addiction. Proc Natl Acad Sci U S A. 1998 Aug 4;95(16):9608-13. doi: 10.1073/pnas.95.16.9608. PMID 9689128
- [Background] Grosch S, Niederberger E, Lotsch J, Skarke C, Geisslinger G. A rapid screening method for a single nucleotide polymorphism (SNP) in the human MOR gene. Br J Clin Pharmacol. 2001 Dec;52(6):711-4. doi: 10.1046/j.0306-5251.2001.01504.x. PMID 11736886
- [Background] Hollt V. A polymorphism (A118G) in the mu-opioid receptor gene affects the response to morphine-6-glucuronide in humans. Pharmacogenetics. 2002 Jan;12(1):1-2. doi: 10.1097/00008571-200201000-00001. No abstract available. PMID 11773858
- [Background] Lotsch J, Skarke C, Grosch S, Darimont J, Schmidt H, Geisslinger G. The polymorphism A118G of the human mu-opioid receptor gene decreases the pupil constrictory effect of morphine-6-glucuronide but not that of morphine. Pharmacogenetics. 2002 Jan;12(1):3-9. doi: 10.1097/00008571-200201000-00002. PMID 11773859
- [Background] LaForge KS, Shick V, Spangler R, Proudnikov D, Yuferov V, Lysov Y, Mirzabekov A, Kreek MJ. Detection of single nucleotide polymorphisms of the human mu opioid receptor gene by hybridization or single nucleotide extension on custom oligonucleotide gelpad microchips: potential in studies of addiction. Am J Med Genet. 2000 Oct 9;96(5):604-15. doi: 10.1002/1096-8628(20001009)96:53.0.co;2-f. PMID 11054767
- [Background] Wang D, Quillan JM, Winans K, Lucas JL, Sadee W. Single nucleotide polymorphisms in the human mu opioid receptor gene alter basal G protein coupling and calmodulin binding. J Biol Chem. 2001 Sep 14;276(37):34624-30. doi: 10.1074/jbc.M104083200. Epub 2001 Jul 16. PMID 11457836
- [Background] Town T, Abdullah L, Crawford F, Schinka J, Ordorica PI, Francis E, Hughes P, Duara R, Mullan M. Association of a functional mu-opioid receptor allele (+118A) with alcohol dependency. Am J Med Genet. 1999 Oct 15;88(5):458-61. PMID 10490697
- [Background] Shi J, Hui L, Xu Y, Wang F, Huang W, Hu G. Sequence variations in the mu-opioid receptor gene (OPRM1) associated with human addiction to heroin. Hum Mutat. 2002 Apr;19(4):459-60. doi: 10.1002/humu.9026. PMID 11933204
- [Background] Schinka JA, Town T, Abdullah L, Crawford FC, Ordorica PI, Francis E, Hughes P, Graves AB, Mortimer JA, Mullan M. A functional polymorphism within the mu-opioid receptor gene and risk for abuse of alcohol and other substances. Mol Psychiatry. 2002;7(2):224-8. doi: 10.1038/sj.mp.4000951. PMID 11840318
- [Background] Sander T, Gscheidel N, Wendel B, Samochowiec J, Smolka M, Rommelspacher H, Schmidt LG, Hoehe MR. Human mu-opioid receptor variation and alcohol dependence. Alcohol Clin Exp Res. 1998 Dec;22(9):2108-10. PMID 9884158
- [Background] Wong CA: Combined spinal-epidural labor analgesia. Techniques in Regional Anesthesia and Pain Management 2003; 7: 181-88
- [Background] Palmer CM, Cork RC, Hays R, Van Maren G, Alves D. The dose-response relation of intrathecal fentanyl for labor analgesia. Anesthesiology. 1998 Feb;88(2):355-61. doi: 10.1097/00000542-199802000-00014. PMID 9477056
- [Background] Nelson KE, Rauch T, Terebuh V, D'Angelo R. A comparison of intrathecal fentanyl and sufentanil for labor analgesia. Anesthesiology. 2002 May;96(5):1070-3. doi: 10.1097/00000542-200205000-00007. PMID 11981144
- [Background] Clarke VT, Smiley RM, Finster M. Uterine hyperactivity after intrathecal injection of fentanyl for analgesia during labor: a cause of fetal bradycardia? Anesthesiology. 1994 Oct;81(4):1083. doi: 10.1097/00000542-199410000-00041. No abstract available. PMID 7943823
- [Background] Landau R, Cahana A, Smiley RM, Antonarakis SE, Blouin JL. Genetic variability of mu-opioid receptor in an obstetric population. Anesthesiology. 2004 Apr;100(4):1030-3. doi: 10.1097/00000542-200404000-00042. No abstract available. PMID 15087647
- [Background] Palmer CM, Emerson S, Volgoropolous D, Alves D. Dose-response relationship of intrathecal morphine for postcesarean analgesia. Anesthesiology. 1999 Feb;90(2):437-44. doi: 10.1097/00000542-199902000-00018. PMID 9952150
- [Background] Ronaghi M, Uhlen M, Nyren P. A sequencing method based on real-time pyrophosphate. Science. 1998 Jul 17;281(5375):363, 365. doi: 10.1126/science.281.5375.363. No abstract available. PMID 9705713
- [Background] Wasson J, Skolnick G, Love-Gregory L, Permutt MA. Assessing allele frequencies of single nucleotide polymorphisms in DNA pools by pyrosequencing technology. Biotechniques. 2002 May;32(5):1144-6, 1148, 1150 passim. doi: 10.2144/02325dd04. PMID 12019788
- [Background] Neve B, Froguel P, Corset L, Vaillant E, Vatin V, Boutin P. Rapid SNP allele frequency determination in genomic DNA pools by pyrosequencing. Biotechniques. 2002 May;32(5):1138-42. doi: 10.2144/02325dd03. PMID 12019787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Laboring subject recruited from 10/2005 to 9/2006 Post cesarean delivery subjects recruited from 10/2005 to 5/2007
Pre-assignment Details: Subjects were excluded from the labor analgesia group if they had received an opioid analgesic before initiation of intrathecal analgesia or if they received neuraxial analgesia before 2cm of cervical dilation.
Groups:
- Labor Analgesia OPRM1 c304A: Parturients that received spinal fentanyl 15 micrograms and epidural fentanyl labor analgesia who were homozygous for OPRM1 c304
- Labor Analgesia OPRM1 c304A>G: Parturients receiving spinal fentanyl 15 micrograms and epidural fentanyl labor analgesia that were heterozygous or homozygous for OPRM1 c304A>G
- Cesarean Delivery OPRM1 c304A: Cesarean delivery subjects receiving morphine 150 micrograms with spinal bupivacaine 12mg and fentanyl 15 micrograms that were homozygous for OPRM1 c304A
- Cesarean Delivery OPRM1 c304A>G: Cesarean delivery subjects receiving morphine 150 micrograms with spinal bupivacaine 12mg and fentanyl 15 micrograms that were heterozygous for OPRM1 c304A>G
Period: Overall Study
Arm/Group | Labor Analgesia OPRM1 c304A | Labor Analgesia OPRM1 c304A>G | Cesarean Delivery OPRM1 c304A | Cesarean Delivery OPRM1 c304A>G
Started | 144 | 46 | 78 | 25
Completed | 144 | 46 | 78 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Labor Analgesia OPRM1 c304A | Labor Analgesia OPRM1 c304A>G | Cesarean Delivery OPRM1 c304A | Cesarean Delivery OPRM1 c304A>G | Total
Number analyzed (Participants) | 144 | 46 | 78 | 25 | 293
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 144 | 46 | 78 | 25 | 293
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [28 to 34] | 32 [30 to 34] | 34 [31 to 37] | 32 [29 to 35] | 32 [28 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 46 | 78 | 25 | 293
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 144 | 46 | 78 | 25 | 293

OUTCOME MEASURES:

1. Primary Outcome: Duration of Intrathecal Fentanyl Analgesia
Description: Time from intrathecal drug administration to request for analgesia either in laboring women of after cesarean delivery
Time Frame: Time (0-1440 minutes) to first analgesia request
Population: Laboring parturients that received intrathecal fentanyl (25 micrograms) for initiation of labor analgesia were evaluated for this outcome per protocol.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Labor Analgesia OPRM1 c304A | Labor Analgesia OPRM1 c304A>G | Cesarean Delivery OPRM1 c304A | Cesarean Delivery OPRM1 c304A>G
Number analyzed (Participants) | 144 | 46 | 0 | 0
Minutes | 70 [62 to 78] | 63 [50 to 76] |  |
Statistical Analysis 1: Comparison: Labor Analgesia OPRM1 c304A vs Labor Analgesia OPRM1 c304A>G; Log rank test; Test type: Superiority or Other; p = 0.54, Log Rank

2. Primary Outcome: Duration of Intrathecal Analgesia Following Cesarean Delivery
Description: Time until request for supplemental analgesia following intrathecal morphine/fentanyl for cesarean delivery
Time Frame: 0 to 72 hours following cesarean delivery
Population: Subjects that received fentanyl and morphine for postpartum analgesia after planned cesarean delivery were analyzed per protocol.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Labor Analgesia OPRM1 c304A | Labor Analgesia OPRM1 c304A>G | Cesarean Delivery OPRM1 c304A | Cesarean Delivery OPRM1 c304A>G
Number analyzed (Participants) | 0 | 0 | 78 | 25
Hours |  |  | 26 [0 to 47] | 40 [0 to 60]
Statistical Analysis 1: Comparison: Cesarean Delivery OPRM1 c304A vs Cesarean Delivery OPRM1 c304A>G; Test type: Superiority or Other; p = 0.15, Log Rank

3. Secondary Outcome: Severity of Pruritus Following Fentanyl
Description: Severity of pruritus during labor analgesia
Time Frame: Labor analgesia
Measure: Number; unit: participants
Arm/Group | Labor Analgesia OPRM1 c304A | Labor Analgesia OPRM1 c304A>G | Cesarean Delivery OPRM1 c304A | Cesarean Delivery OPRM1 c304A>G
Number analyzed (Participants) | 144 | 46 | 0 | 0
participants
  None | 9 | 13 |  |
  Mild | 48 | 59 |  |
  Moderate | 35 | 26 |  |
  Severe | 8 | 2 |  |
Statistical Analysis 1: Comparison: Labor Analgesia OPRM1 c304A vs Labor Analgesia OPRM1 c304A>G; Test type: Superiority or Other; p = 0.06, Chi-squared, Corrected

4. Secondary Outcome: Subjects With Pruritus at 24 Hours Post Morphine
Description: Subjects reporting pruritus in the first 24 hours post cesarean delivery
Time Frame: 24 hours post cesarean delivery
Measure: Number; unit: participants
Arm/Group | Labor Analgesia OPRM1 c304A | Labor Analgesia OPRM1 c304A>G | Cesarean Delivery OPRM1 c304A | Cesarean Delivery OPRM1 c304A>G
Number analyzed (Participants) | 0 | 0 | 78 | 25
participants |  |  | 33 | 3
Statistical Analysis 1: Comparison: Cesarean Delivery OPRM1 c304A vs Cesarean Delivery OPRM1 c304A>G; Test type: Superiority or Other; p = 0.02, Chi-squared, Corrected

5. Primary Outcome: Visual Analog Pain Scale (0 to 100) at Analgesia Request Following Intrathecal Intervention
Description: Visual analog pain scale (0 to 100) at 1st request for supplemental analgesia
Time Frame: VAS at analgesia request
Population: Analysis population per protocol.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Labor Analgesia OPRM1 c304A | Labor Analgesia OPRM1 c304A>G | Cesarean Delivery OPRM1 c304A | Cesarean Delivery OPRM1 c304A>G
Number analyzed (Participants) | 144 | 46 | 78 | 25
Units on a scale | 33 [21 to 50] | 38 [23 to 51] | 26 [0 to 47] | 40 [0 to 60]
Statistical Analysis 1: Comparison: Labor Analgesia OPRM1 c304A vs Labor Analgesia OPRM1 c304A>G; Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cesarean Delivery OPRM1 c304A vs Cesarean Delivery OPRM1 c304A>G; Test type: Superiority or Other; p = 0.84, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Labor Analgesia OPRM1 c304A | Labor Analgesia OPRM1 c304A>G | Cesarean Delivery OPRM1 c304A | Cesarean Delivery OPRM1 c304A>G
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/46 | 0/78 | 0/25
Other Adverse Events (participants affected / at risk) | 0/144 | 0/46 | 0/78 | 0/25

LIMITATIONS AND CAVEATS:
A limitation to the finding of this study was the relatively low number of OPRM1 heterozygous subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No